CLINICAL TRIAL: NCT03293290
Title: Project EMPOWERING: Evidence-based PrEP for Justice-Involved Women and Their Risk Networks
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1606017882
Record Dates: First submitted 2017-09-20; First posted 2017-09-26 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: HIV Infections
Keywords: HIV pre-exposure prophylaxis; criminal justice; women; risk networks
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- PrEP (Experimental): For participants who are eligible for PrEP and willing to participate, subjects on PrEP will be followed for 1 year with quarterly assessments.
  Interventions: Drug: PrEP

INTERVENTIONS:
Drug: PrEP — Subjects on PrEP will be followed for 1 year with quarterly assessments by trained research assistants. Study visits will take place at in New Haven and Hartford. At every scheduled visit, participants will receive a comprehensive package of preventive services, including a prescription for the next 30-day supply of TDF/FTC (with 2 refills), a symptom screen for acute HIV, risk-reduction counseling, PrEP adherence support, bleach for cleaning injection equipment, and condoms. HIV rapid testing with Orasure® will be performed quarterly; participants testing newly positive for HIV (representing seroconversions) will be followed with confirmatory testing and referred to care as needed.
  Other Names: TDF/FTC

SUMMARY:
This study has two components. The first component is designed to assess and compare the awareness, attitudes and clinical eligibility of Pre-exposure Prophylaxis (PrEP) in criminal justice (CJ) involved women. The second component is designed to evaluate the acceptability and feasibility of strategically delivering PrEP to CJ involved women and their risk network members.

DETAILED DESCRIPTION:
Risk networks can be leveraged to maximally disseminate effective interventions to women, including PrEP, and thereby potentially avert some of the 50,000 annual incident HIV infections in the U.S. Few studies to date have capitalized on risk networks as a way to identify and engage high-risk individuals, like CJ-involved women, who could markedly benefit from PrEP. This study advances the field by: 1) Using an innovative network-based framework (a non-traditional model of care delivery) to engage a high risk population in PrEP dissemination as HIV prevention; 2) Incorporating a syndemic approach to PrEP that addresses HIV prevention in the context of substance use, psychiatric comorbidities, IPV, and stigma; and 3) Recruiting, enrolling, and retaining high risk networks of CJ-involved women who are difficult to reach by other means. In doing so, this proposal addresses key funding priorities of the Gilead Investigator Sponsored Research program, which includes research on PrEP implementation targeted to high risk populations and delivered in non-traditional clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* Index participants reside in, or planning to reside in New Haven or Hartford, Connecticut,.
* Criminal justice-involved (anticipate release or have been released from prison or jail within 6 months, and/or are under or anticipating transfer to correctional community supervision (i.e. probation or parole)).
* Self-reported HIV negative.

Eligible and enrolled women will then recruit risk network members through respondent driven sampling, using vouchers.

Risk network members must:

* have a unique and valid referral coupon (from Index participant).
* Reside or planning to reside in New Haven or Hartford, Connecticut.
* Self-reported HIV negative
* 18 years of age or older

Exclusion Criteria:

* They are unable or unwilling to provide informed consent.
* Are threatening to staff.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Cis- or trans- female participants are eligible.
Enrollment: 105 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
% PrEP uptake | Month 1
  # starting PrEP/ # enrolled subjects
% eligible PrEP uptake | Month 1
  # starting PrEP/ # eligible subjects

SECONDARY OUTCOMES:
Mean % PrEP adherence | 12 months
  # PrEP pills taken/# PrEP pills prescribed per month
Mean TDF level | 12 months
  TDF level by dried blood spot testing
HIV incidence | 12 months
  New HIV+ by 4th generation HIV Ag/Ab testing

CONTACTS AND LOCATIONS:
Overall Officials: Jaimie Meyer, MD, MS, FACP, Principal Investigator — Yale University
Locations (1):
- Yale Clinical and Community Research, 270 Congress Ave, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Meyer JP, Price CR, Ye Y, Qin Y, Tracey D, Demidont AC, Melbourne K, Altice FL. A PrEP Demonstration Project Using eHealth and Community Outreach to Justice-Involved Cisgender Women and Their Risk Networks. AIDS Behav. 2022 Dec;26(12):3807-3817. doi: 10.1007/s10461-022-03709-2. Epub 2022 Jun 7. PMID 35672552